CLINICAL TRIAL: NCT03151746
Title: Effect of Preoperative Gabapentin on Postoperative Pain Associated With Ureteroscopy and Stents Insertion: a Double Blind, Randomized, Placebo Controlled Trial
Brief Title: Gabapentin on Postoperative Pain Associated With Ureteroscopy and Stents Insertion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Luminita M. Tureanu, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00205047
Record Dates: First submitted 2017-04-19; First posted 2017-05-12 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia; Urethral Obstruction
MeSH Terms: conditions — Urethral Obstruction | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Double Blind, Randomized, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded by using placebo or active drug supplied by Investigational Drug Pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo pill administered 1 hour before planned surgical procedure
  Interventions: Drug: Placebo
- Gabapentin (Experimental): Gabapentin pill (1200mg) administered orally 1 hour prior to planned surgical procedure
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Placebo — Placebo pill administered orally 1 hour before planned surgical procedure
  Arms: Placebo
Drug: Gabapentin — Gabapentin pill (1200mg) administered orally 1 hour before planned surgical procedure
  Arms: Gabapentin

SUMMARY:
The study's objective is to determine the efficacy of preoperative gabapentin in relieving postoperative pain, reducing opioid use and improving quality of recovery in subjects undergoing urologic surgery.

Investigators hypothesize that subjects receiving gabapentin will have lower pain scores, less opioid consumption and better quality of recovery as compared to subjects who are given a placebo.

DETAILED DESCRIPTION:
Approximately one hour prior to induction of anesthesia in preoperative holding area all enrolled subjects will receive PO Acetaminophen 650 mg, the Gabapentin group will receive PO Gabapentin 1200 mg, while the Control group will receive PO Placebo, with a small amount of water.

Upon arrival in the operating room, standard ASA monitors will be applied. Intraoperative, patients will receive a standardized anesthetic care. This care consists of induction with IV propofol 2mg/kg, IV fentanyl 2 mcg/kg (adjusted body weight), and IV rocuronium 0.6 mg/kg for tracheal intubation or IV succinylcholine 1mg/kg if rapid sequence induction is needed.

For maintenance of general anesthesia, investigators will use Sevoflurane, with the goal to maintain BP within 20% of preoperative baseline and BIS 40-60.

If HR > 100/min and BIS 40-60 may use IV esmolol 0.5 mg/kg. If BP and/or HR >20% preoperative baseline, and BIS 40- 60 despite above management, may titrate IV antihypertensive agents.

For PONV prophylaxis, 30 min before end of surgery investigatorswill administer IV ondansetron 8mg.

The time from end of surgery to extubation in OR will be documented with a free text note in the EMR.

After extubation all patients will be transported to PACU on 2-liter Oxygen by nasal cannula, which will be weaned off in the PACU.

The postoperative analgesics during Phase I of recovery in PACU will consist of IV Hydromorphone 0.2-0.4 mg prn pain to maintain adequate pain control (NPRS<4). During Phase II of recovery patients will receive PO Hydromorphone 2mg tablets every 4-6 hours as needed for pain (NPRS ≥ 4) and acetaminophen: 650mg PO every 6 hours

The following data will be collected every hour during phase I and phase II recovery:

* pain (NPRS)
* sedation (Ramsey sedation scale)
* dizziness (1- mild, 2- moderate, 3- severe)
* headache YES/No If yes: NPRS score HA
* respiratory depression (hypoventilation/ apnea: RR < 10 bpm., desaturation: (SpO2 < 90%)
* Sedated but still in pain (Yes/No)
* PONV YES/NO
* PONV receiving antiemetic treatment
* time to first opioid administration (IV hydromorphone)
* total amount of IV hydromorphone in PACU Phase I
* total amount of oral analgesic (hydromorphone) in PACU Phase II
* time to meet discharge criteria from PACU Phase I
* time to meet discharge criteria from Phase II

Study research personnel will contact participants by phone or in the hospital at 24 hours and 48 hours postoperative and at approximately one week in the Urology clinic. The study research personnel will ask questions regarding pain (NPRS) and analgesic consumption. The IPSS and QOR-40 questionnaires will be administered and data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 75 years
* Patients with obstructive kidney stones undergoing elective ureteroscopy or cystoscopy with Ureteral stent placement

Exclusion Criteria:

* Age less than 18 or more than 75 years
* Acetaminophen allergy
* Gabapentin allergy
* Hydromorphone allergy
* Chronic use of gabapentin
* History of chronic pain (Pain for > than 3 months)
* Chronic renal insufficiency (Creatinine > 1.3)
* Seizure disorder
* Psychiatric disorders (medically treated)
* Chronic use of anticonvulsants, antidepressants, antipsychotics (use > 3 months)
* Antacids ingested within 2 hours prior to surgery
* History of gastric or duodenal ulcer
* Pregnant or lactating
* Inability to communicate in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luminita Tureanu, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi HB, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG, Barry MJ. Indwelling ureteral stents: evaluation of symptoms, quality of life and utility. J Urol. 2003 Mar;169(3):1065-9; discussion 1069. doi: 10.1097/01.ju.0000048980.33855.90. PMID 12576847
- [Background] Koprowski C, Kim C, Modi PK, Elsamra SE. Ureteral Stent-Associated Pain: A Review. J Endourol. 2016 Jul;30(7):744-53. doi: 10.1089/end.2016.0129. Epub 2016 May 23. PMID 27125392
- [Background] Schmidt PC, Ruchelli G, Mackey SC, Carroll IR. Perioperative gabapentinoids: choice of agent, dose, timing, and effects on chronic postsurgical pain. Anesthesiology. 2013 Nov;119(5):1215-21. doi: 10.1097/ALN.0b013e3182a9a896. No abstract available. PMID 24051389
- [Background] Mason CJ. High frequency jet ventilation through a Robertshaw double lumen tube. Anaesthesia. 1986 Mar;41(3):330. doi: 10.1111/j.1365-2044.1986.tb12811.x. No abstract available. PMID 3963344
- [Background] Bala I, Bharti N, Chaubey VK, Mandal AK. Efficacy of gabapentin for prevention of postoperative catheter-related bladder discomfort in patients undergoing transurethral resection of bladder tumor. Urology. 2012 Apr;79(4):853-7. doi: 10.1016/j.urology.2011.11.050. Epub 2012 Feb 4. PMID 22309784

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Gabapentin
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gabapentin | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (16.4) | 49 (14.72) | 49 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 7 | 10 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20
Height (Inches) [Mean (Standard Deviation); unit: Inches] | 67.2 (3.27) | 67.7 (4.33) | 67.5 (3.89)
Weight (kilograms) [Mean (Standard Deviation); unit: Kilograms] | 89.58 (21.6) | 76.1 (17.48) | 83.4 (19.74)

OUTCOME MEASURES:

1. Primary Outcome: 48 Hours Morphine Equivalents Consumed.
Description: Total morphine equivalents in milligrams consumed during the first 48 hours after surgery.
Time Frame: Up to 48 hours after surgery
Measure: Mean (Full Range); unit: morphine milligrams
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 9 | 11
morphine milligrams | 51.87 [0 to 204] | 15.71 [0 to 48]

2. Secondary Outcome: 24 Hour Pain Burden
Description: Pain scores using an 11 point numeric pain rating scale 0=no pain 10 = worst pain imaginable
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 9 | 11
score on a scale | 4.11 (2.26) | 3.11 (2.67)

3. Secondary Outcome: QOR 40 Questionnaire Scores
Description: Evaluate quality of recovery using the Quality of Recovery 40 (QoR 40) questionnaire a 40 question survey scored from 40 ( poor recovery) to 200 high (good recovery) 48 hours after the surgical procedure.
Time Frame: 48 hours after surgical procedure
Population: 3 in the placebo and 3 in the gabapentin group did not complete the survey at 48 hours post operative.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 6 | 8
score on a scale | 181.3 [160 to 198] | 187.5 [171 to 200]

ADVERSE EVENTS:
Time Frame: 7 days after surgical procedure.
Arm/Group | Placebo | Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 2/9 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Gabapentin (N=11)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Headache (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (11) — Headache
Dizziness (General disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The limitation to this study is that enrollment was affected by COVID 19 protocols within the hospital enrollment. This is why the project was terminated early .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03151746/Prot_SAP_000.pdf